CLINICAL TRIAL: NCT03497988
Title: Effect of a Single Dose of Intranasal Oxytocin on Food Intake in Obese Adolescents
Brief Title: Intranasal Oxytocin and Food Intake in Obese Adolescents
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Grant proposal not funded, study has been withdrawn with IRB
Sponsor: Shana McCormack, MD (Other)
Responsible Party: Sponsor-Investigator, Shana McCormack, MD, Attending Physician, Sponsor Investigator, Children's Hospital of Philadelphia
Organization: Children's Hospital of Philadelphia (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 17-014360
Record Dates: First submitted 2018-03-19; First posted 2018-04-13 (Actual); Last update posted 2018-12-26 (Actual); Status verified 2018-12

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Syntocinon (=Oxytocin), then Placebo (Experimental): 1. Single-Dose Intranasal Oxytocin
  2. Single-Dose Placebo
  Interventions: Drug: Syntocinon; Drug: Placebo
- Placebo, then Syntocinon (=Oxytocin) (Experimental): 1. Single-Dose Placebo
  2. Single-Dose Intranasal Oxytocin
  Interventions: Drug: Syntocinon; Drug: Placebo

INTERVENTIONS:
Drug: Syntocinon — The active substance of Syntocinon is a synthetic nonapeptide identical to the posterior pituitary hormone oxytocin.
  Other Names: Intranasal Oxytocin
Drug: Placebo — The placebo is identical to the Syntocinon formulation with the exception of the active compound, i.e., without oxytocin.
  Other Names: Placebo (for Syntocinon)

SUMMARY:
The purpose of the study is to determine the effect of intranasal OXT caloric intake and eating behaviors in otherwise healthy obese adolescents.

The primary objective of this study is to determine the effects of intranasal administration of oxytocin on food intake in obese, pubertal or post-pubertal adolescents (13 to <18 years in girls, and 15 to <20 years in boys).

DETAILED DESCRIPTION:
Participants will undergo a telephone screening and then, within 4 weeks, complete an in-person screening visit to determine eligibility. Then, within 4 weeks they will be randomized to either OXT or placebo. After a minimum 1-week (7-28 days) "washout," participants will cross-over to treatment with the other condition (i.e., placebo or OXT).

ELIGIBILITY:
Inclusion Criteria:

1. Proficient in English.
2. Pubertal or Post-Pubertal Females: 13 to <18 years.
3. Pubertal or Post-Pubertal Males: 15 to <20 years.
4. Girls must have a negative urine pregnancy test and post-menarchal girls must use an acceptable method of contraception, including abstinence, a barrier method (diaphragm or condom), Depo-Provera, or an oral contraceptive, for the duration of the study.
5. Currently obese (BMI >95%ile for age/sex if age < 18 years, BMI > 30 kg/m2 age 18 - 20 years). In children, obesity is defined with respect to age- and sex based as greater than or equal to the 95th%ile1, whereas in adults, an absolute threshold is used.
6. Parental/guardian permission (informed consent) and if appropriate, child assent.

Exclusion Criteria:

1. Diabetes mellitus requiring insulin or insulin secretagogue. (Laboratory values: HgbA1c ≥8.5%)
2. Cardiovascular condition, as defined as any of the following: i) abnormal blood pressure, defined as <3%ile or >97%ile for age, sex and height 3, for adult participants abnormal blood pressure is defined as Stage 2 hypertension (systolic BP > 160 mm Hg or diastolic BP > 100 mm Hg); ii) history of cardiac arrhythmia or arrhythmia detected on screening ECG; iii) history of heart failure and/or cardiomyopathy; iv) prolonged QTc interval (QTc > 460 msec), and/or long QT syndrome phenotype and/or positive genotype for long QT syndrome pathogenic mutations.
3. Concurrent use of medications known to prolong QTc interval and pose high risk for Torsades de Pointes (TdP) according to the current information available (www.crediblemeds.org). Concomitant medications will be assessed by the Investigational Drug Service (IDS) pharmacist, in collaboration with the study cardiologist, if additional clarification is needed. In addition, we require that potential participants be on a stable dose for at least 2 months of any medication with the potential to alter cardiac rhythm to ensure the screening ECG reflects steady-state physiology.
4. Laboratory abnormalities that indicate abnormal sodium level, liver or renal disease, or anemia:

   Sodium - Outside Normal Range; Aspartate Aminotransferase (AST)/SGOT > 3.0 X's Upper Limit of Normal (ULN); Alanine Aminotransferase (ALT)/SGPT > 3.0 X's Upper Limit of Normal (ULN); Estimated Glomerular Filtration Rate (eGFR) < 60 mL/min/1.73m2; Hemoglobin < 10 g/dL
5. Seizure in the past 12 mos.
6. History of gastrectomy, gastric bypass, small or large bowel resection.
7. History of active substance abuse.
8. Current use of psychiatric medications. Current psychotic disorder and/or suicidality.
9. Other chronic medical conditions or medications likely to affect appetite or food intake.
10. Any investigational drug use within 30 days prior to enrollment.
11. Pregnant or lactating females.
12. Inability to take intranasal medication (e.g., recent injury)
13. Parents/guardians or subjects who, in the opinion of the Investigator, may be non-compliant with study schedules or procedures.

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2018-09 (Estimated); Primary Completion 2020-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Effect on Food Intake | 28 Days
  Kilocalories Consumed at as desired ('Ad Lib') Test Meal

SECONDARY OUTCOMES:
Adverse Events | 28 Days
  Number of participants with adverse events.
Effect of OXT on Eating Behaviors at Mealtime (appetite) | 28 Days
  Investigators will assess appetite, a visual analog scale (VAS) to quantify participants' self-reported appetite on a linear scale will be used. The range of the VAS is 0% to 100% of the scale, with 0% corresponding to no self-reported appetite, and 100% corresponding to maximal self-reported appetite.
Effect of OXT on Eating Behaviors at Mealtime (impulsivity) | 28 Days
  Investigators will measure impulsivity, which may affect the decision to eat, performance on a computerized stop-signal task will be assessed. Outcome measures include: direction errors (#, more = more errors), proportion of successful stops (%, higher = more successful), reaction time on "Go" trials (longer = slower), stop signal reaction time (longer= slower).

CONTACTS AND LOCATIONS:
Overall Officials: Shana E McCormack, MD, MTR, Principal Investigator — Children's Hospital of Philadelphia

IPD SHARING:
Plan to Share IPD: No